CLINICAL TRIAL: NCT00298337
Title: Use of Probiotic Bacteria in Prevention of Allergic Disease in Children 1999-2008
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Helsinki (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: T101060058;T1040A0002;T110612
Record Dates: First submitted 2006-03-01; First posted 2006-03-02 (Estimated); Last update posted 2006-10-18 (Estimated); Status verified 2006-03

CONDITIONS: Atopic Dermatitis; Food Hypersensitivity; Allergic Rhinitis, Seasonal; Allergic Conjunctivitis; Asthma
MeSH Terms: conditions — Dermatitis, Atopic; Food Hypersensitivity; Rhinitis, Allergic, Seasonal; Conjunctivitis, Allergic; Asthma

INTERVENTIONS:
Drug: Mixture of probiotic bacteria and prebiotic oligosaccharide

SUMMARY:
The aim of the study is to find out if allergic diseases can be prevented buy giving probiotic bacteria to pregnant mothers and their newborn infants

ELIGIBILITY:
Inclusion Criteria:

* mother or father fo child with doctor diagnoses allergic disease

Exclusion Criteria:

* prematurity, major malformations

Ages: 37 Weeks to 42 Weeks | Sex: All
Age Groups: Child
Dates: Start 1999-10; Study Completion 2007-12

CONTACTS AND LOCATIONS:
Overall Officials: Erkki Savilahti, Professor, Study Chair — Helsinki University Central Hospital, Hospital for Children and Adults, PO Box 281, 00029 HUS, Finland
Locations (1):
- Helsinki University Central Hospital, Skin and Allergy Hospital, Helsinki, PO Box 160, Finland

REFERENCES:
- [Derived] Kallio S, Jian C, Korpela K, Kukkonen AK, Salonen A, Savilahti E, Kuitunen M, M de Vos W. Early-life gut microbiota associates with allergic rhinitis during 13-year follow-up in a Finnish probiotic intervention cohort. Microbiol Spectr. 2024 Jun 4;12(6):e0413523. doi: 10.1128/spectrum.04135-23. Epub 2024 Apr 30. PMID 38687061
- [Derived] Tarrant I, Finlay BB. Human milk oligosaccharides: potential therapeutic aids for allergic diseases. Trends Immunol. 2023 Aug;44(8):644-661. doi: 10.1016/j.it.2023.06.003. Epub 2023 Jul 11. PMID 37438187
- [Derived] Korpela K, Kallio S, Salonen A, Hero M, Kukkonen AK, Miettinen PJ, Savilahti E, Kohva E, Kariola L, Suutela M, Tarkkanen A, de Vos WM, Raivio T, Kuitunen M. Gut microbiota develop towards an adult profile in a sex-specific manner during puberty. Sci Rep. 2021 Dec 2;11(1):23297. doi: 10.1038/s41598-021-02375-z. PMID 34857814
- [Derived] Kallio S, Kukkonen AK, Savilahti E, Kuitunen M. Perinatal probiotic intervention prevented allergic disease in a Caesarean-delivered subgroup at 13-year follow-up. Clin Exp Allergy. 2019 Apr;49(4):506-515. doi: 10.1111/cea.13321. Epub 2018 Dec 18. PMID 30472801
- [Derived] Korpela K, Salonen A, Vepsalainen O, Suomalainen M, Kolmeder C, Varjosalo M, Miettinen S, Kukkonen K, Savilahti E, Kuitunen M, de Vos WM. Probiotic supplementation restores normal microbiota composition and function in antibiotic-treated and in caesarean-born infants. Microbiome. 2018 Oct 16;6(1):182. doi: 10.1186/s40168-018-0567-4. PMID 30326954
- [Derived] Savilahti EM, Kukkonen AK, Haahtela T, Tuure T, Kuitunen M, Savilahti E. Intestinal defensin secretion in infancy is associated with the emergence of sensitization and atopic dermatitis. Clin Exp Allergy. 2012 Mar;42(3):405-11. doi: 10.1111/j.1365-2222.2011.03904.x. Epub 2011 Nov 16. PMID 22093109
- [Derived] Kukkonen AK, Savilahti EM, Haahtela T, Savilahti E, Kuitunen M. Ovalbumin-specific immunoglobulins A and G levels at age 2 years are associated with the occurrence of atopic disorders. Clin Exp Allergy. 2011 Oct;41(10):1414-21. doi: 10.1111/j.1365-2222.2011.03821.x. Epub 2011 Jul 19. PMID 21771118
- [Derived] Kukkonen K, Savilahti E, Haahtela T, Juntunen-Backman K, Korpela R, Poussa T, Tuure T, Kuitunen M. Long-term safety and impact on infection rates of postnatal probiotic and prebiotic (synbiotic) treatment: randomized, double-blind, placebo-controlled trial. Pediatrics. 2008 Jul;122(1):8-12. doi: 10.1542/peds.2007-1192. PMID 18595980
- See also: Clinical trials — http://www.hus.fi